CLINICAL TRIAL: NCT04708288
Title: A PROSPECTIVE, MULTI-CENTER, SINGLE-ARM, POST MARKET OBSERVATIONAL STUDY TO EVALUATE THE SAFETY AND CLINICAL PERFORMANCE OF THE ARCHIMEDES BIODEGRADABLE BILIARY AND PANCREATIC STENT
Acronym: AM GI Registry
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: QualiMed Innovative Medizinprodukte GmbH (Industry)
Responsible Party: Sponsor
Other Study IDs: 2680
Record Dates: First submitted 2021-01-08; First posted 2021-01-13 (Actual); Last update posted 2023-03-29 (Actual); Status verified 2023-03

CONDITIONS: Obstructed Biliary and Pancreatic Duct

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: ARCHIMEDES Biodegradable Biliary and Pancreatic Stent — Pts that will receive ARCHIMEDES Biodegradable Biliary and Pancreatic Stent

SUMMARY:
Significant experience with biodegradable materials has been reported in the orthopedic literature; in particular; biodegradable stents have been used in the endovascular and urologic epithelium. Stents are typically made from polymeric materials including Polylactic Acid (PLA), Polyglycolide (PGA), Polydioxanone (PDO), Polyethyleneglycol (PEG), Polycaprolactone (PCL), etc., which have been cleared or approved by the FDA and CE-marked as drug carriers, sutures, and bone fixatives. The material is degraded by hydrolysis in, e.g., lactic acid, which is removed from the body by normal metabolic pathways. In the field of gastroenterology, these stents were first introduced in patients with an esophageal stenosis with encouraging results, although esophageal hyperplasia was a frequently encountered complication.

For biliary applications, biodegradable stents have been evaluated in several in-vitro and animal studies that demonstrated that the stents were safe and well tolerated. These stents provided an adequate radial force and resulted in complete stricture resolution within several months. The stents did not show any signs of biliary hyperplasia or integration in the epithelium. Moreover, they seem to have a self-clearing effect on attached biofilm as the outer layer sloughs during the degradation process similarly to the exfoliation of human skin. Also, the stent could be removed from the bile duct, thus offering the possibility of extraction if necessary at various times after implantation.

In 2010, Petryl was the first to use a biodegradable stent in the human bile duct. A stent was successfully placed using percutaneous transhepatic cholangiograpy in two patients with a postsurgical intrahepatic biliary stricture. Transient cholangitis was the only complication encountered and during the two years of follow-up, the bile duct remained patent.

Later, Mauri et al. presented in 2013 and 2016 results of a 107 patient study on a polydioxanone biodegradable biliary stent. The results have been published in the Journal of the European Society of Radiology. The authors concluded that percutaneous placement of a biodegradable biliary stent is a feasible and safe strategy to treat benign biliary strictures refractory to standard bilioplasty, with promising results in the mid-term period.

Prior to this study, the ARCHIMEDES device was assessed in the ARCHIMEDES Investigational study which has completed enrolment with 53 patients included, and the results are not yet published. In this study approximately half the stents were deployed in the bile duct (53%) and half in the pancreatic duct. All 53 patients have either completed, exited, or no longer have the study device. No patient remains in the study with a stent in place during the time of the last patient follow-ups. The study concluded without any device-related SAE. Bilirubin was reduced by 25.6%, which exceeded the >20% clinical success criterion, quality of life score improved from 3.7 to 7.9, procedural success was rated 1.4 (good to excellent), and technical success was achieved in all 53 patients.

Data from the ARCHIMEDES Investigational study was used for CE Mark approval, which was obtained in June 2018.

ELIGIBILITY:
Inclusion Criteria:

* Patient eligible for implantation of a pancreatic or billiary stent prior to participate in the study and according to current guidelines
* Patient has provided a signed and dated informed consent (according to the laws and regualtions of the country in which the observational study is conducted)

Exclusion Criteria:

* Age < 18 y
* Inability to understand the purpose of the study or refusal to cooperate
* Not available for routine follow-up visits
* Pregnancy
* Currently participating in a confounding trial before reaching first endpoint.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients that will respect the inlcusion criteria will be enrolled in the study.
Sampling Method: Non-Probability Sample
Enrollment: 198 (Estimated)
Dates: Start 2020-09-22 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Safety data of the procedure | 24 months
  Number of patients with adverse events
Clinical performance of the procedure | 24 months
  Number of patients with better synthomatology

CONTACTS AND LOCATIONS:
Locations (8):
- HUS Helsinki University Hospital, Helsinki, Finland
- Evangelisches Krankenhaus Düsseldorf, Düsseldorf, Germany
- Emek Medical Center, Afula, Israel
- Italy (3):
  - Endoscopy Unit, Humanitas Research Hospital, Rozzano, Milano
  - AUSL Romagna Ospedale Morgagni - Pierantoni, Forlì
  - UCBM - Campus Bio-Medico University, Roma
- University Medical Center Ljubljana, Ljubljana, Slovenia
- Hospital Universitario de Salamanca, Salamanca, Spain

IPD SHARING:
Plan to Share IPD: No